CLINICAL TRIAL: NCT04598529
Title: Impact of A2 Milk Versus Conventional Milk on Intestinal Health: a Proof-of-concept Study in Irritable Bowel Syndrome Patients
Brief Title: Impact of A2 Milk Versus Conventional Milk on Intestinal Health: a Proof-of-concept Study in IBS-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NL73898.068.20; METC 20-032 (Other: Medical Ethical Committee)
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; IBS-C; IBS-D; Conventional milk; A2 milk; Gastrointestinal symptoms
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A2 milk (Active Comparator): A2 milk, organic, 200ml, twice daily
  Interventions: Other: A2 milk
- Conventional milk (Placebo Comparator): Pasteurized semi-skimmed milk, organic, 200ml, twice daily
  Interventions: Other: Conventional milk

INTERVENTIONS:
Other: A2 milk — a variety of cow's milk that contains only A2 beta-casein (and therefore lacks of A1 beta-casein).
  Arms: A2 milk
Other: Conventional milk — cow's milk with a mixture of A1 and A2 beta-casein.
  Arms: Conventional milk

SUMMARY:
This aim of this study is to evaluate the acute and mid-term effects of A2 milk versus conventional milk on gastrointestinal symptoms in patients with constipation-predominant IBS and in patients with diarrhea-predominant IBS. Moreover, the effect of immune and defense markers will be studied.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a prevalent functional bowel disorder in which recurrent abdominal pain is associated with defecation and altered bowel habits. Although the pathophysiology is incompletely understood, it is generally regarded as a multifactorial disorder involving host factors such as low-grade immune activation, altered intestinal barrier function and defense. Environmental factors, including diet, are also suggested to play a role. Dairy products such as cow's milk are widely produced and an important component of the human diet. Cow's milk is composed of various macronutrients, micronutrients and water. Beta-casein is a major protein component of cow's milk; most cows produce a mixture of A1 and A2 beta-casein (conventional milk), whereas some cows produce only A2 beta-casein (A2 milk). It has been suggested that specific components in cow's milk, such as A1 beta-casein, may trigger gastrointestinal symptoms after intake.

The purpose of this randomized, double-blind, cross-over study performed in Maastricht University Medical Center (MUMC+) is to explore the acute and mid-terms effects of A2 milk versus conventional milk on gastrointestinal symptoms and immune and defense markers in separate groups of patient with constipation-predominant IBS and in patients with diarrhea-predominant IBS.

ELIGIBILITY:
Inclusion Criteria:

* IBS with constipation (IBS-C) or IBS with diarrhea (IBS-D), based on the Rome IV criteria
* Self-reported indication that dietary components (e.g. milk) trigger GI symptoms
* Body Mass Index (BMI) < 30 kg/m2
* Weight-stable for at least 90 days prior to participation (no change in bodyweight, i.e. < 3kg).
* Willing to be informed in case of unexpected findings.

Exclusion Criteria:

* History of any disease or surgery interfering with the study aims, limiting participating or completing the study protocol
* Self-admitted human immunodeficiency virus-positive state.
* Disease with a life expectancy shorter than 5 years.
* Abdominal surgery interfering with gastrointestinal function (to be decided by a medical doctor)
* Based on anamnesis, patients with lactose intolerance will be excluded. If not tested before, a lactose breath test can be performed to check for lactose intolerance.
* Self reported cow's milk allergy
* Use of antibiotics within 30 days prior to the study
* Use of other medication interfering with study outcomes, as will be reviewed by a medical doctor, who will decide on in- or exclusion based on the drug(s) used
* Administration of probiotic or prebiotic supplements, investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principle investigator), in the 14 days prior to the study
* Known pregnancy or lactation
* Plan to loose weight or follow a specific diet within the study period
* Alcohol intake: female >7 units/week for females, male >14 units/week
* Blood donation within 1 month prior to the study
* Insufficient fluency of the Dutch language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
The acute effects of A2 milk versus conventional milk on overall gastrointestinal discomfort in separate groups of individuals with IBS-C and IBS-D. | On the 1 day intervention period
  Assessed by a single item using a visual analogue scale (VAS), anchored at the low end (score of 0) with the absence of overall symptoms and at the other end (score of 100) with severe symptoms, the worst it has ever been.

SECONDARY OUTCOMES:
The mid-term effects of A2 milk versus conventional milk on overall gastrointestinal discomfort in separate groups of individuals with IBS-C and IBS-D. | up to 3 days (once daily) after 1 day of intervention
  Assessed by a single item using a visual analogue scale (VAS), anchored at the low end (score of 0) with the absence of overall symptoms and at the other end (score of 100) with severe symptoms, the worst it has ever been.
The acute and mid-term effects of A2 milk versus conventional milk on single gastrointestinal symptoms and stool characteristics in separate groups of individuals with IBS-C and IBS-D. | Multiple times at the 1 day intervention day and once daily up to 3 days after intervention day
  Assessed by a visual analogue scale (VAS) for different gastrointestinal symptoms, anchored at the low end (score of 0) with the absence of overall symptoms and at the other end (score of 100) with severe symptoms, the worst it has ever been.
The mid-term effects of A2 milk versus conventional milk on single gastrointestinal symptoms and stool characteristics in separate groups of individuals with IBS-C and IBS-D. | At the first intervention day
  Assessed by the IBS-SSS questionnaire (a 0-100 scale, with the total IBS-SSS score ranging between 0 and 500, with higher scores indicating more severe symptoms).
The mid-term effects of A2 milk versus conventional milk on gastrointestinal immune and defense markers in separate groups of individuals with IBS-C and IBS-D. | At both intervention days
  Assessed by several parameters of GI immune and defense in feces.

CONTACTS AND LOCATIONS:
Overall Officials: D.M.A.E. Jonkers, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Currently, we do not anticipate on sharing data outside MUMC+. If this changes in the future, we will submit an amendment.